CLINICAL TRIAL: NCT00930735
Title: The Prognostic Significance of Fibrosis Detection in Ischemic and Non-ischemic Cardiomyopathy
Brief Title: The Prognostic Significance of Fibrosis Detection in Cardiomyopathy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Sanjay Prasad, Consultant Cardiologist, Royal Brompton & Harefield NHS Foundation Trust
Other Study IDs: 09/0904
Record Dates: First submitted 2009-06-27; First posted 2009-06-30 (Estimated); Last update posted 2018-04-23 (Actual); Status verified 2018-04

CONDITIONS: Cardiomyopathy; Coronary Artery Disease
MeSH Terms: conditions — Cardiomyopathies; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum and plasma and myocardium
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Myocardial fibrosis, outcomes: Groups with none and variable amounts of myocardial fibrosis

SUMMARY:
The presence of scar within heart muscle can act as a substrate for abnormal rhythm problems and lead to the developement of heart failure

Clinical significance Correlation with biomarkers and genetic markers

DETAILED DESCRIPTION:
Patients will undergo cardiovascular magnetic resonance (CMR) to include measurement of left ventricular volumes, ejection fraction, detection of inflammation (via STIR sequences) where appropriate, early gadolinium enhancement, late gadolinium enhancement, first pass perfusion using pharmacological stress imaging (contraindications to include comorbidities that do not permit pharmacological stress agents e.g. severe asthma, severe or symptomatic aortic stenosis)

ELIGIBILITY:
Inclusion Criteria:

* presence of an ischaemic or non-ischaemic cardiomyopathic process
* no contraindication to contrast enhanced CMR
* GFR >30

Exclusion Criteria:

* ESRF
* Contraindication to CM R

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive referrals for CMR from tertiary and nontertiary referral hospitals scanned to evaluate presence and amount of myocardial scarring.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2000-01; Primary Completion 2020-04-30 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
All cause mortality | 3 years
Ventricular arrhythmias | 3 years
Unplanned heart failure admissions | 3 years

SECONDARY OUTCOMES:
Ejection fraction | 3
NYHA status | 3

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay K Prasad, MD, Principal Investigator — Royal Brompton and Harefield Foundation Trust
Locations (1):
- Royal Brompton Hospital, London, United Kingdom

REFERENCES:
- [Derived] Vassiliou VS, Pavlou M, Malley T, Halliday BP, Tsampasian V, Raphael CE, Tse G, Vieira MS, Auger D, Everett R, Chin C, Alpendurada F, Pepper J, Pennell DJ, Newby DE, Jabbour A, Dweck MR, Prasad SK. A novel cardiovascular magnetic resonance risk score for predicting mortality following surgical aortic valve replacement. Sci Rep. 2021 Oct 12;11(1):20183. doi: 10.1038/s41598-021-99788-7. PMID 34642428
- [Derived] Halliday BP, Gulati A, Ali A, Guha K, Newsome S, Arzanauskaite M, Vassiliou VS, Lota A, Izgi C, Tayal U, Khalique Z, Stirrat C, Auger D, Pareek N, Ismail TF, Rosen SD, Vazir A, Alpendurada F, Gregson J, Frenneaux MP, Cowie MR, Cleland JGF, Cook SA, Pennell DJ, Prasad SK. Association Between Midwall Late Gadolinium Enhancement and Sudden Cardiac Death in Patients With Dilated Cardiomyopathy and Mild and Moderate Left Ventricular Systolic Dysfunction. Circulation. 2017 May 30;135(22):2106-2115. doi: 10.1161/CIRCULATIONAHA.116.026910. Epub 2017 Mar 28. PMID 28351901
- [Derived] Dawson DK, Hawlisch K, Prescott G, Roussin I, Di Pietro E, Deac M, Wong J, Frenneaux MP, Pennell DJ, Prasad SK. Prognostic role of CMR in patients presenting with ventricular arrhythmias. JACC Cardiovasc Imaging. 2013 Mar;6(3):335-44. doi: 10.1016/j.jcmg.2012.09.012. Epub 2013 Feb 20. PMID 23433931
- [Derived] Dweck MR, Joshi S, Murigu T, Gulati A, Alpendurada F, Jabbour A, Maceira A, Roussin I, Northridge DB, Kilner PJ, Cook SA, Boon NA, Pepper J, Mohiaddin RH, Newby DE, Pennell DJ, Prasad SK. Left ventricular remodeling and hypertrophy in patients with aortic stenosis: insights from cardiovascular magnetic resonance. J Cardiovasc Magn Reson. 2012 Jul 28;14(1):50. doi: 10.1186/1532-429X-14-50. PMID 22839417
- [Derived] Dweck MR, Joshi S, Murigu T, Alpendurada F, Jabbour A, Melina G, Banya W, Gulati A, Roussin I, Raza S, Prasad NA, Wage R, Quarto C, Angeloni E, Refice S, Sheppard M, Cook SA, Kilner PJ, Pennell DJ, Newby DE, Mohiaddin RH, Pepper J, Prasad SK. Midwall fibrosis is an independent predictor of mortality in patients with aortic stenosis. J Am Coll Cardiol. 2011 Sep 13;58(12):1271-9. doi: 10.1016/j.jacc.2011.03.064. PMID 21903062
- [Derived] O'Hanlon R, Grasso A, Roughton M, Moon JC, Clark S, Wage R, Webb J, Kulkarni M, Dawson D, Sulaibeekh L, Chandrasekaran B, Bucciarelli-Ducci C, Pasquale F, Cowie MR, McKenna WJ, Sheppard MN, Elliott PM, Pennell DJ, Prasad SK. Prognostic significance of myocardial fibrosis in hypertrophic cardiomyopathy. J Am Coll Cardiol. 2010 Sep 7;56(11):867-74. doi: 10.1016/j.jacc.2010.05.010. Epub 2010 Jun 25. PMID 20688032